CLINICAL TRIAL: NCT03055312
Title: A Randomized, Multicenter,Phase III Study of Bicalutamide Versus Chemotherapy in First Line Treatment of AR Positive Metastatic Triple Negative Breast Cancer
Brief Title: Bicalutamide in Treatment of Androgen Receptor (AR) Positive Metastatic Triple Negative Breast Cancer
Acronym: SYSUCC-007
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSUCC-007
Record Dates: First submitted 2017-01-09; First posted 2017-02-16 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Drug Therapy; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TPC chemotherapy (Active Comparator): Conventional chemotherapy(choose a):
  TX (Taxotere and Xeloda),GT (Gemcitabine and Paclitaxel),GC (Gemcitabine and Carboplatin)
  Interventions: Drug: TPC
- Bicalutamide (Experimental): Bicalutamide 150mg/day every 28 days
  Interventions: Drug: Bicalutamide 150 mg

INTERVENTIONS:
Drug: TPC — Conventional chemotherapy(choose a):
  TX:(Docetaxel 75mg/m2 iv day1 and Capecitabine 950mg/m2 po twice daily days 1-14)every 3 weeks.
  GT:(Paclitaxel 175mg/m2 iv day1 and Gemcitabine 1250mg/m2 iv days 1 & days 8)every 3 weeks.
  GC:(Gemcitabine 1000mg/m2 on days 1 & days 8 and Carboplatin by Area Under Curve (AUC) 2 iv on days 1 & days 8) every 3 weeks
  Other Names: Chemotherapy
  Arms: TPC chemotherapy
Drug: Bicalutamide 150 mg — Bicalutamide 150mg/day,every 28 days
  Other Names: Bicalutamide
  Arms: Bicalutamide

SUMMARY:
Compare the efficacy of bicalutamide with conventional chemotherapy (Treatment of Physician's Choice,TPC) in first-line treatment of AR positive metastatic triple negative breast

DETAILED DESCRIPTION:
This is a phase III,Multi-center,prospective,randomized clinical trials. The objective compare the efficacy of bicalutamide with conventional chemotherapy (Treatment of Physician's Choice,TPC) in first-line treatment of AR positive metastatic triple negative breast cancer.Primary endpoint is 16-week clinical benefit rate (CBR).By centre randomized grouping bicalutamide (experimental Group) or TPC (Control Group).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old, female
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Confirmed by pathology or organizing cytology AR positive(IHC：≧10%)triple negative breast cancer
* For the first time recurrence or newly diagnosed advanced breast cancer,Disease-free survival time 12 months above
* Measurable disease per RECIST version 1.1,or immeasurably lesions bone metastasis
* After Recurrence has not received cancer treatment
* Life expectancy of at least 6 months
* Signed and dated an informed consent form

Exclusion Criteria:

* ECOG score ≧2
* Only brain metastasis or meningeal metastasis
* Receiving other anti-tumor treatment
* Heart,lung,liver,kidney,bone marrow,and other functions badness

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate for 16 weeks | 16 weeks
  The proportion of patients with complete response, partial response and stable disease

SECONDARY OUTCOMES:
progression-free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Yuan, M.D, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No